CLINICAL TRIAL: NCT06829797
Title: A Multicenter Randomized Controlled Phase II Trial of Iparomlimab and Tuvonralimab (QL1706) Combined with SOX Chemotherapy Versus Chemotherapy Alone in the Treatment of Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma(STAR-03)
Brief Title: A Multicenter Randomized Controlled Phase II Trial of Iparomlimab and Tuvonralimab (QL1706) Combined with SOX Chemotherapy Versus Chemotherapy Alone in the Treatment of Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: STAR-03
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Li Leping, Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.2024-1046
Record Dates: First submitted 2025-02-06; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QL1706+SOX group (Experimental)
  Interventions: Drug: Neoadjuvant Therapy(QL1706+SOX Chemotherapy); Procedure: Radical surgery (D2); Drug: Drug: Adjuvant therapy(QL1706+SOX chemotherapy)
- SOX group (Active Comparator)
  Interventions: Drug: Neoadjuvant Therapy(SOX Chemotherapy); Procedure: Radical surgery (D2); Drug: Drug: Adjuvant therapy(SOX chemotherapy)

INTERVENTIONS:
Drug: Neoadjuvant Therapy(QL1706+SOX Chemotherapy) — Preoperative QL1706 combined with SOX regimen (4 cycles) → Radical surgery (D2) → Postoperative QL1706 combined with SOX regimen (4 cycles). QL1706 (50mg/2mL) , at a dose of 5mg/kg, the desired volume of drug is withdrawn and slowly infused into an IV bag of 0.9% NaCl, prepared as a diluent with a final concentration of 1-10mg/mL, mixed, and infused intravenously, Q3W, administered on the first day of each cycle.
  Arms: QL1706+SOX group
Drug: Neoadjuvant Therapy(SOX Chemotherapy) — Preoperative SOX regimen (4 cycles) → radical surgery (D2) → postoperative SOX regimen (4 cycles).
  Arms: SOX group
Procedure: Radical surgery (D2) — Surgical treatment is completed within 3-5 weeks after the end of neoadjuvant therapy.
Drug: Drug: Adjuvant therapy(QL1706+SOX chemotherapy) — Postoperative adjuvant therapy is 4 cycles of QL1706+SOX chemotherapy.
  Arms: QL1706+SOX group
Drug: Drug: Adjuvant therapy(SOX chemotherapy) — Postoperative adjuvant therapy is 4 cycles of SOX chemotherapy.
  Arms: SOX group

SUMMARY:
To explore the efficacy of Iparomlimab and Tuvonralimab (QL1706) in combination with SOX chemotherapy versus chemotherapy alone for the neoadjuvant treatment of locally-progressed gastric/gastroesophageal union adenocarcinomas by evaluating the complete pathologic remission rate (pCR).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study and signing of informed consent;
* Age ≥18 years and ≤75 years;
* Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma;
* Clinical staging of T3N+ or T4a any N, M0 (according to AJCC 8th edition staging), with potential radical resection confirmed by CT or MRI;
* Have not received any anti-tumor therapy (e.g., surgery, radiotherapy, chemotherapy, targeted therapy and immunotherapy);
* Planned to undergo surgery after completion of neoadjuvant therapy;
* Be able to swallow pills normally;
* ECOG-PS score 0-1;
* Expected survival ≥ 12 months;
* Normal major organ function.

Exclusion Criteria:

* Known HER2 positivity;
* Known peritoneal metastases or positive peritoneal cytology (CY1P0) or T4b (according to AJCC 8th edition);
* Presence of unresectable factors including unresectable tumors, contraindications to surgery and refusal of surgery;
* The presence of a pre-existing or concurrent malignancy, with the exception of cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and carcinoma in situ of the breast
* History of gastrointestinal perforation, history of abdominal abscess or recent (within 3 months) occurrence of intestinal obstruction, or concomitant intestinal obstruction as indicated by imaging or clinical signs;
* Patients with abnormal coagulation (International Normalized Ratio (INR) >2.0 or Prothrombin Time (PT) >16s), a bleeding tendency or currently receiving thrombolytic or anticoagulant therapy (prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed);
* Clinically significant bleeding symptoms or significant bleeding tendency such as gastrointestinal bleeding, gastric ulcer bleeding, and vasculitis within 3 months prior to randomization into groups. Patients with positive fecal occult blood at baseline may be retested, and if the retest remains positive, gastroscopy will be required (except for patients who have had a gastroscopy within 3 months prior to enrollment to rule out this condition);
* Arterial/venous thrombotic events such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, and cerebral infarction), deep vein thrombosis, and pulmonary embolism within 6 months prior to randomization to group;
* A known hereditary or acquired predisposition to bleeding and thrombosis (e.g., hemophilia, coagulation disorders, and thrombocytopenia);
* The presence of active ulcers, unhealed wounds or fractures
* Urinalysis showing urinary protein ≥++, confirmed by 24-hour urine protein quantification >1.0 g;
* Active infections requiring antimicrobial therapy (e.g., antibacterial, antiviral, and antifungal medications);
* Active hepatitis (Hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/mL; Hepatitis C reference: HCV antibody positive and HCV viral copy number > upper limit of normal (ULN));
* Congenital or acquired immunodeficiency (e.g., HIV-infected patients);
* Planned or previous organ or allogeneic bone marrow transplant;
* Current interstitial pneumonia or interstitial lung disease, or a history of interstitial pneumonia or interstitial lung disease requiring hormonal therapy, or other conditions that may interfere with the assessment and management of immune-related pulmonary toxicity, such as pulmonary fibrosis, opportunistic pneumonia (e.g., occlusive bronchiectasis), pneumoconiosis, drug-associated pneumonia, and idiopathic pneumonitis, or active pneumonitis or severe pulmonary impairment as demonstrated by CT at screening; Active tuberculosis;
* Any active autoimmune disease or history of autoimmune disease with potential for relapse;
* Treatment with immunosuppressive drugs or systemic corticosteroids (>10 mg/day of prednisone or equivalent) within 7 days prior to randomization to group;
* Use of a strong CYP3A4 inducer within 2 weeks prior to randomization subgroup or use of a strong CYP3A4 inhibitor within 1 week prior to randomization subgroup
* Oral or intravenous administration of therapeutic antibiotics within 4 weeks prior to randomization to subgroups, except for prophylactic antibiotics administered intravenously for no more than 48 hours
* Known allergy to any study drug or excipient;
* Participation in a clinical study of another drug within 4 weeks prior to randomization to group;
* Being a lactating female.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 14-16 weeks.
  Pathological complete response was defined as pT0N0M0

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 14-16 weeks.
  The percentage of surviving tumor cells in the tumor bed after neoadjuvant therapy was ≤10%.
R0 resection rate | From date of neoadjuvant therapy until the date of postoperative pathological assessment, assessed up to 14-16 weeks.
  The proportion of patients who completed R0 resection in the total enrolled patients.
Event-free survival (EFS) | From date of neoadjuvant therapy until the date of the first occurrence of the above events, assessed up to 60 months.
  From the beginning of the study to the time of the first occurrence of any of the following events, disease progression beyond surgical treatment, local or distant recurrence, death from any cause, etc.
Overall survival (OS) | From the date of diagnosis to the date of death, assessed up to 60 months.
  From study inception to patient death from any cause.
Disease-free survival (DFS) | From date of neoadjuvant therapy until the date of the disease recurrence or death due to disease progression, assessed up to 60 months.
  The time from randomization until disease recurrence or death due to disease progression.
Surgical safety | From date of neoadjuvant therapy until the date of 30 days post-surgery, assessed up to 17-19 weeks.
  The occurrence of postoperative complications including surgical site infection, anastomotic leakage, gastrointestinal bleeding, incisional dehiscence, adhesive bowel obstruction, biliary and celiac fistulae, and unexplained fever (≥37.5°C).
Adverse Events | From the date of neoadjuvant therapy to the completion of postoperative adjuvant therapy, up to 24 months.
  Based on NCI-CTCAE (version 5.0) adverse events (AEs): including type, incidence, grading, severity, duration, and relevance to the study drug
Drug tolerance | From the date of neoadjuvant therapy to the completion of postoperative adjuvant therapy, up to 24-28 weeks.
  The proportion of dose interruptions, dose reductions, and discontinuations due to drug-related toxicity during the study period.
Prognostic Biomarkers | From the date of neoadjuvant therapy initiation until the end of postoperative follow-up, up to 24 months.
  Biomarkers of interest include PD-L1 expression (assessed by IHC), microsatellite instability (MSI) status (determined by PCR-based testing), tumor mutation burden (TMB) (evaluated using next-generation sequencing), and circulating tumor DNA (ctDNA) levels (quantified via liquid biopsy). The correlation between these biomarkers and treatment efficacy, including progression-free survival (PFS) and overall survival (OS), will be analyzed.

IPD SHARING:
Plan to Share IPD: Undecided